CLINICAL TRIAL: NCT05797545
Title: Comparison of Ultrasound and Breast MRI for Breast Cancer Detection Among Women With Dense Breasts and a Personal History of Breast Cancer
Brief Title: Comparison of Ultrasound and Breast MRI for Breast Cancer Detection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Eun Sook Ko, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2022-11-076-002
Record Dates: First submitted 2023-02-22; First posted 2023-04-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Mass Screening; Ultrasonography; Magnetic Resonance Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abbreviated Breast MRI for Breast Cancer Detection (Experimental): Women are classified and randomly assigned into MRI sequence groups(1st round screening/2nd round screening : AB (abbreviated)-MRI / FP (full protocol)-MRI application group and FP (full protocol)-MRI / AB (abbreviated)). MRI (either AB-MRI or FP-MRI) assigned as the 1st round screening (baseline), mammography, and ultrasound are performed on the same day. For the 2nd round screening one year after the 1st round screening, a different MRI (i.e., FP-MRI if AB-MRI was performed in the previous year, AB-MRI if FP-MRI was performed in the previous year), mammography, and ultrasound were performed on the same day as the 1st round screening.
  Interventions: Diagnostic Test: Breast MRI for Breast Cancer Detection
- Full Protocol MRI for Breast Cancer Detection (Experimental): Women are classified and randomly assigned into MRI sequence groups(1st round screening/2nd round screening : AB (abbreviated)-MRI / FP (full protocol)-MRI application group and FP (full protocol)-MRI / AB (abbreviated)). MRI (either AB-MRI or FP-MRI) assigned as the 1st round screening (baseline), mammography, and ultrasound are performed on the same day. For the 2nd round screening one year after the 1st round screening, a different MRI (i.e., FP-MRI if AB-MRI was performed in the previous year, AB-MRI if FP-MRI was performed in the previous year), mammography, and ultrasound were performed on the same day as the 1st round screening.
  Interventions: Diagnostic Test: Breast MRI for Breast Cancer Detection

INTERVENTIONS:
Diagnostic Test: Breast MRI for Breast Cancer Detection — Comparison of diagnostic results of abbreviated breast MRI and full protocol MRI for secondary breast cancer surveillance

SUMMARY:
The goal of this randomized clinical trial is to compare diagnostic results of secondary breast cancer surveillance using breast ultrasound abbreviated MRI and full protocol MRI.

DETAILED DESCRIPTION:
Women who have been treated for breast cancer are at risk of ipsilateral local/regional recurrence or new primary cancers in the contralateral breast, which are associated with increased rates of distant metastases and breast cancer mortality. The goal of post-treatment imaging surveillance is to detect early second breast cancer, which permits interventions to improve survival and maintain quality of life.

Currently, most guidelines consistently recommend annual mammography for women with a personal history of breast cancer (PHBC). However, in women with dense breasts, mammographic sensitivity decreased from a level of 85.7%-88.8% in patients with almost entirely fatty tissue to 62.2%-68.1%. Even more, sensitivity of mammography was lower in women with a PHBC within the initial 5 years after primary breast cancer (PBC) treatment. In addition, dense breasts lead to an increased percentage of interval cancer. Thus, the need for a better surveillance modality has emerged.

In this context, breast US may be considered as a supplemental screening modality because it is widely available, does not need contrast agents, and is of relatively lower cost . A few studies indicate that adding screening US to mammography reduced interval cancer rates for women with dense breasts and enable detection of early-stage cancers at an average of 4.2 cancers per 1000 US examinations. As an another candidate, breast MRI shows high sensitivity and offers the highest cancer detection rate but its routine usage in women with a PHBC is still on debate.

Another possible imaging modality is breast magnetic resonance imaging (MRI). Current National Comprehensive Cancer Network (NCCN) guidelines suggest annual screening with mammography and MRI is recommended for ① women with Breast Cancer Susceptibility Gene (BRCA1 or BRCA2) mutations, ② first-degree family members of carriers of BRCA mutations, ③ women with a lifetime risk of breast cancer greater than 20% based on family history, and ④ women have radiotherapy for thorax at the age of 10-30 years and ⑤ women diagnosed with lobular carcinoma in situ (LCIS), atypical ductal hyperplasia (ADH), or atypical lobular hyperplasia (ALH) by previous biopsy. And, this is based on the results of existing single-center or multi-center prospective studies. Women who underwent breast-conserving surgery for breast cancer before the age of 50 were added to the 2018 new MRI screening group of the American College of Radiology (ACR), and their secondary breast cancer risk is 20% or more. Most women with a history of breast cancer have an intermediate risk (>15% but <20%) of developing breast cancer. Therefore, when most patients are not in the high-risk group, performing conventional MRI (full-protocol MRI, FP-MRI) for all postoperative examinations is not appropriate in terms of cost and time.

Abbreviated MRI (AB-MRI), introduced relatively recently, is a method designed to increase accessibility by reducing time and cost by selectively capturing only some sequences in FP-MRI. Sequence composition can be adjusted in various ways, and image acquisition must be completed within 10 minutes. A number of studies have demonstrated that AB-MRI has comparable diagnostic results to FP-MRI. The most recent paper published in Korea compared the scores of 726 patients with AB-MRI and FP-MRI by performing propensity score matching. The results were comparable in sensitivity, and AB-MR was significantly higher in specificity. Other indicators such as interval cancer rate or Breast Imaging Reporting & Data System (BI-RADS) Category 3 rate did not show significant differences between the two groups. However, all studies are retrospective and there are no prospective data. Since the reported scores of AB-MRI and FP-MRI are comparable, it is difficult to test because the sample size is larger than 18,000 in order to perform a non-inferiority test on diagnostic scores. The purpose of this study was to compare the diagnostic results of secondary breast cancer surveillance using mammography, ultrasound, and MRI in a prospective multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-75 with a history of breast cancer (in situ carcinoma or invasive breast cancer [stage 0-3])
* Women with dense breasts with pattern C (heterogeneously dense) or D (extremely dense breasts) using AI-based Lunit INSIGHT for Mammography (version 1.1.4.3, Lunit Inc.) in the most recent mammography
* Women who have not had a breast imaging test within 6 months
* Women who agreed to undergo regular annual mammography, breast ultrasound, and breast MRI

Exclusion Criteria:

* Patients with symptoms related to current breast cancer or breast cancer recurrence (palpable mass, bloody or transparent nipple secretion, palpable mass in the axillary region, abnormal skin changes in the breast or nipple)
* If you have been diagnosed with regional recurrence (axillary lymph nodes, supraclavicular and subclavian lymph nodes, internal mammary lymph nodes, etc.) or distant metastases
* In case of bilateral total mastectomy
* If women are receiving chemotherapy for cancer in other organs
* Women during pregnancy or lactation
* Glomerular filtration rate < 30 mL/min/1.73m2, or patients with renal insufficiency on dialysis
* If women have severe claustrophobia
* If women have a metal prosthesis that is not suitable for MR (e.g. breast tissue expander, etc.)
* If there is a history of severe contrast agent side effects (e.g., anaphylactoid reaction, dyspnea, etc.)

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1756 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2028-05-28 (Estimated); Study Completion 2028-05-28 (Estimated)

PRIMARY OUTCOMES:
Cancer detection rate (CDR) | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of cancer detection rate (CDR) between breast ultrasound and abbreviated magnetic resonance imaging (AB-MRI) or breast ultrasound and full protocol magnetic resonance imaging (FP-MRI)

SECONDARY OUTCOMES:
Abnormal interpretation rate (AIR) | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of abnormal interpretation rate in each test (mammography, ultrasound, abbreviated magnetic resonance imaging (AB-MRI), and full protocol magnetic resonance imaging (FP-MRI))
Sensitivity | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of sensitivity of each test (mammography, ultrasound, abbreviated magnetic resonance imaging (AB-MRI), and full protocol magnetic resonance imaging (FP-MRI))
Specificity | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of specificity of each test (mammography, ultrasound, abbreviated magnetic resonance imaging (AB-MRI), and full protocol magnetic resonance imaging (FP-MRI))
Positive predictive value | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of positive predictive value of each test (mammography, ultrasound, abbreviated magnetic resonance imaging (AB-MRI), and full protocol magnetic resonance imaging (FP-MRI))
Negative predictive value | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of negative predictive value of each test (mammography, ultrasound, abbreviated magnetic resonance imaging (AB-MRI), and full protocol magnetic resonance imaging (FP-MRI))
Interval cancer rate | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Interval cancer rate will be assessed for each test (mammography, ultrasound, abbreviated magnetic resonance imaging (AB-MRI), and full protocol magnetic resonance imaging (FP-MRI))
Invasive cancer detection rate | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of invasive cancer detection rate between breast ultrasound and abbreviated magnetic resonance imaging (AB-MRI) or breast ultrasound and full protocol magnetic resonance imaging (FP-MRI)
Accuracy | The results of pathology tests or imaging or clinical follow-up tests 1 year after the 2nd round screening were used.
  Comparison of accuracy between breast ultrasound and abbreviated magnetic resonance imaging (AB-MRI) or breast ultrasound and full protocol magnetic resonance imaging (FP-MRI)
Patient reported outcomes (PRO) based on patient discomfort. | Patient questionnaires will be collected at time points of clinic visits for study, assessed up to 3 months.
  To compare patient reported outcome related to diagnostic testing with AB-MR and full-protocol MR based on patient discomfort. This dimension is rated on a 5-point scale from 1 (no problem) to 5 (extreme problems).
Patient reported outcomes (PRO) based on patient preference. | Patient questionnaires will be collected at time points of clinic visits for study, assessed up to 3 months.
  To compare patient reported outcome related to diagnostic testing with AB-MR and full-protocol MR based on patient preference. This dimension is rated on a 5-point scale from 1(AB-MR is twice as preferable as FP-MR) to 5(FP-MR is twice as preferable as AB-MR).

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sook Ko, M.D., Ph.D., Study Chair — Samsung Medical Center; Yung Mi Park, M.D., Ph.D., Principal Investigator — Inje University; Yun woo Jang, M.D., Ph.D., Principal Investigator — Soon Chun Hyang University
Locations (3):
- South Korea (3):
  - Inje University Busan Paik Hospital, Busan, BusanJin-Gu
  - Samsung Medical center, Seoul, Gangnam-gu
  - Soon Chun Hyang University Hospital Seoul, Seoul, Yongsan-Gu

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: date relative to the time when summary data are published or otherwise made available (for example, starting 6 months after publication
Access Criteria: The study chair and principle investigators will review requests and criteria for reviewing requests

REFERENCES:
- [Derived] Chang YW, Park YM, Kim K, Kim MJ, Kim MK, Yu J, Ko ES. Prospective Multicenter Study Comparing Magnetic Resonance Imaging and Ultrasonography for Second Breast Cancer Surveillance in Women With Prior Breast Cancer and Dense Breasts: KBCSG-27 Trial. J Breast Cancer. 2025 Dec;28(6):427-436. doi: 10.4048/jbc.2025.0121. Epub 2025 Oct 23. PMID 41311334